CLINICAL TRIAL: NCT03785574
Title: Study of Different Therapeutic Strategies in Hydatidiform Mole With Lung Nodule，A Prospective Multicentre Randomized Controlled Trial
Brief Title: Study of Different Therapeutic Strategies in Hydatidiform Mole With Lung Nodule
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Tongji Hospital Affiliated to Tongji Medical College of HUST (Unknown); The First People's Hospital of Yunnan (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); Women and Children's Hospital of Ningbo University (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Hangzhou Fuyang Women And Children Hospital (Unknown); Zhejiang Provincial Tongde Hospital (Other); Shaoxing Shangyu Women And Children Hospital (Unknown); Huzhou Maternity and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Lixiao, Professor, Women's Hospital School Of Medicine Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSEM 012
Record Dates: First submitted 2018-12-21; First posted 2018-12-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hydatidiform Mole; Gestational Trophoblastic Neoplasia
Keywords: Pulmonary Nodule; Chemotherapy; Chorionic Gonadotrophin
MeSH Terms: conditions — Hydatidiform Mole; Gestational Trophoblastic Disease | interventions — Drug Therapy; Methotrexate

STUDY DESIGN:
Intervention Model Description: lung nodule ≥1.0cm were randomized into 2 groups: A. treated with chemotherapy immediately, B. follow up until hCG level met FIGO diagnostic criteria of GTN (B1) or hCG level declined to normal spontaneously (B2). A:B=1:2，the sample size of group A and group B was 30 in total.
  Lung nodule <1.0cm will be directly treated as group C: follow up until hCG level met FIGO diagnostic criteria of GTN (C1) or hCG level declined to normal spontaneously (C2), it is an observation study and the sample volume depends on the enrolling time of group A and B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A:chemotherapy immediately (Active Comparator): Treated with chemotherapy immediately. First line treatments：low risk：Methotrexate or ACTD; high risk：EMA-CO
  Interventions: Drug: chemotherapy
- B:follow up (Experimental): B1: follow up until hCG level met FIGO diagnostic criteria of GTN, then chemotherapy.
  B2: follow up until hCG level declined to normal spontaneously.
  Interventions: Other: Follow up; Drug: chemotherapy
- C: lung nodule diameter <1.0 cm (Experimental): C1: follow up until hCG level met FIGO diagnostic criteria of GTN, then chemotherapy. C2: follow up until hCG level declined to normal spontaneously.
  Interventions: Other: Follow up; Drug: chemotherapy

INTERVENTIONS:
Other: Follow up — the follow up group would be naturely didived into 2 subgroups depending the hCG regression degree.
  Other Names: not chemotherapy immediately
  Arms: B:follow up; C: lung nodule diameter <1.0 cm
Drug: chemotherapy — First line treatments：low risk：Methotrexate or ACTD; high risk：EMA-CO
  Other Names: mtx for low risk

SUMMARY:
The purpose of present study is to provide clinical evidences for the appropriate management of molar pregnancy with lung nodule. The hydatidiform mole patients with lung nodule ≥1.0cm will be randomized into 2 groups: A. treated with chemotherapy immediately, B. follow up until hCG level met FIGO diagnostic criteria of GTN (B1) or hCG level declined to normal spontaneously (B2). Lung nodule <1.0cm will directly treated as group C

DETAILED DESCRIPTION:
The hydatidiform mole patients with lung nodule ≥1.0cm will be randomized into 2 groups: A. treated with chemotherapy immediately, B. follow up until hCG level met FIGO diagnostic criteria of GTN (B1) or hCG level declined to normal spontaneously (B2). The clinical characteristics of patients were compared, especially chemotherapy cycles to achieve hCG normalization and failure to first-line chemotherapy.

Lung nodule <1.0cm will directly treated as group C: follow up until hCG level met FIGO diagnostic criteria of GTN (C1) or hCG level declined to normal spontaneously (C2)

ELIGIBILITY:
Inclusion criteria

Eligible patients have to meet all of the following criteria:

1. Pathologically confirmed HM.
2. The lung nodules are detected by lung CT and metastatic lesions could not be excluded (before or after the suction dilation and curettage).
3. The hCG level does not meet FIGO diagnostic criteria (2018) of GTN.
4. The patients are willing to compliant with the study protocol and be followed up at regular intervals.
5. The patients agree to sign an informed consent form.

Exclusion criteria

1. The patients with a previous history of lung nodules.
2. The imaging impression of lung nodules suggested definitely caused by other diseases, such as tuberculosis, pneumonia, etc.
3. The patients have undergone prophylactic hysterectomy or chemotherapy.
4. Pathologically confirmed gestational trophoblastic neoplasia before and at enrollment.
5. Patients have immunosuppressive diseases or take immunosuppressants.
6. Patients are participating in other clinical trials at same time.
7. Patients were unable or unwilling to provide written informed consent.

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
chemotherapy cycles | 120 months
  the efficacy and number of treatment cycles in the chemotherapy group
hCG declined to normal spontaneously of group B | 120 months
  the spontaneous regression rate in Group B

SECONDARY OUTCOMES:
follow up of group A , B and C | 240 months
  the proportion of spontaneous regression in the follow-up groups, progression-free survival (PFS) and overall survival (OS) in the chemotherapy group
lung nodules | 240 months
  the changes of lung nodules

CONTACTS AND LOCATIONS:
Overall Officials: Xing Xie, Principal Investigator — Women's Hospital, Zhejiang University School of Medicine
Locations (1):
- Weiguo Lv, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No